CLINICAL TRIAL: NCT06235060
Title: The Effect of Two Dıfferent Technıques Used in Psychomotor Skılls Traınıng on Self-Confıdence And Anxıety in Clınıcal Decısıon-Makıng and Academıc Success of Nursıng Students: A Randomızed Controlled Trıal
Brief Title: The Effect of Two Dıfferent Technıques Used in Psychomotor Skılls Traınıng on Nursıng Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ozlem Sahin Akboga, ASSISTANT PROFESSOR, Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CAST
Record Dates: First submitted 2024-01-15; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Anxiety; Clinical Decision-making; Simulation Training; Nursing Students
Keywords: Anxiety; Clinical decision-making; Simulation training; Nursing students
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It is an experimental study with a pretest-posttest design with two intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAST GROUP (Experimental): After the training given with the demonstration method, the training videos on https://www.montgomerycollege.edu/academics/departments/nursing-tpss/nursing-simulation-scenario-library.html were shown to the participants using interactive training methods in parallel with this training. Each session lasted approximately 30-45 minutes. The sessions were repeated in the same environment on the same day and time, once a week, for a total of four weeks (four times).
  Interventions: Other: Computer-assisted simulation technique training group
- Imagery GROUP (Experimental): After the training given with the demonstration method, scenarios suitable for the imagery technique were prepared by the second trainer (Ö.S.A.) in parallel with this training and CAST training. The internal mental visualization format (as if the students were doing the events themselves) was preferred for the imagery technique. The content of the scenarios was examined by three academic nurses who completed their doctoral education in addition to the authors, and expert opinions were taken. The flow of the scenarios was discussed with the experts until a consensus was reached and the final scenario was created. This technique lasted approximately 30-35 minutes.
  Interventions: Other: Imagery GROUP

INTERVENTIONS:
Other: Computer-assisted simulation technique training group — After the training given with the demonstration method, the training videos on https://www.montgomerycollege.edu/academics/departments/nursing-tpss/nursing-simulation-scenario-library.html were shown to the participants using interactive training methods in parallel with this training.
  Other Names: CAST GROUP
  Arms: CAST GROUP
Other: Imagery GROUP — After the training given with the demonstration method, scenarios suitable for the imagery technique were prepared by the second trainer (Ö.S.A.) in parallel with this training and CAST training.
  Other Names: Imagery technique group
  Arms: Imagery GROUP

SUMMARY:
Background: Nursing education aims to provide students with knowledge and skills related to the profession and develop students in terms of personal characteristics such as clinical decision-making, problem-solving, and critical thinking. Innovative approaches and interactive learning strategies are needed during education periods to increase skills and personal development.

Aim: The study aimed to investigate the effect of computer simulation and imagery learning techniques in psychomotor skills training of nursing students on self-confidence and anxiety in clinical decision-making and academic achievement.

Design: It is an experimental study with a pretest-posttest design with two intervention groups.

Setting: The study was conducted between December 2023 and January 2024 at the faculty of health sciences of a university in Turkey's central region.

DETAILED DESCRIPTION:
Background: Nursing education aims to provide students with knowledge and skills related to the profession and develop students in terms of personal characteristics such as clinical decision-making, problem-solving, and critical thinking. Innovative approaches and interactive learning strategies are needed during education periods to increase skills and personal development.

Aim: The study aimed to investigate the effect of computer simulation and imagery learning techniques in psychomotor skills training of nursing students on self-confidence and anxiety in clinical decision-making and academic achievement.

Design: It is an experimental study with a pretest-posttest design with two intervention groups.

Setting: The study was conducted between December 2023 and January 2024 at the faculty of health sciences of a university in Turkey's central region.

Methods: The Turkish version of the "Self-Confidence and Anxiety in Clinical Decision Making" scale was used at the beginning (pre-test) and end (post-test) of the four-week sessions of the interventions. Moreover, the "Academic Achievement Test" was used at the end of the interventions. Differences in mean scores between the groups were analyzed with mixed-design ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* taking the Fundamentals of Nursing course for the first time,
* being have to attend to the Fundamentals of Nursing course,
* having a GPA above 1.80,
* volunteering to participate in the study. It was determined that there were 96 students enrolled in the Fundamentals of Nursing course.

Exclusion Criteria:

* who did not attend regularly during the sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Primer Outcome | PRE TEST-POST TEST (1 month apart)
  Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale: It was developed by White et al. in 2011. The Turkish validity and reliability study of the scale was performed by Bektaş et al. (2017). The scale consists of two sections (self-confidence and anxiety) and 27 items on a six-point Likert scale. The scale has three sub-dimensions for both self-confidence and anxiety sections; "using sources to acquire information and listening to them carefully (13 questions)", "using the information in hand to determine the problem (7 questions)", and "knowing and taking action (7 questions)". Separate scores are obtained for self-confidence and anxiety. As the score obtained from the self-confidence section increases, students' self-confidence levels increase. As the score obtained from the anxiety section decreases, students' anxiety levels decrease. The lowest score that can be obtained from the self-confidence and anxiety sections is 27, and the highest score is 162.

SECONDARY OUTCOMES:
Secondary Outcome | post test (after 1 month)
  Academic Achievement Test: This test was prepared by the researchers. The test included a total of 20 questions related to the subjects taught. A minimum of 0 points and a maximum of 100 points can be obtained from the test. The higher the score obtained from the test, the higher the level of success.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Yozgat Bozok Univercity, Yozgat
  - Yozgat Bozok Universıty, Yozgat

IPD SHARING:
Plan to Share IPD: No